CLINICAL TRIAL: NCT05500235
Title: Scaling Up Tobacco Control in Lndia: Comparing Smartphone to In-person Training for Implementing an Evidence-based Intervention to Reduce Tobacco Use Among Schoolteachers
Brief Title: Comparing Smartphone to In-person Training to Scale Up a Tobacco Control Program for Teachers in India
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Healis-Sekhsaria Institute for Public Health (Other)
Responsible Party: Principal Investigator, Eve Nagler, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB20-2157; R01CA248910-01A1 (NIH)
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-06

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smart phone based training (Experimental): Smartphone-based training for Headmasters to implement the Tobacco Free Teachers-Tobacco Free Society program in their schools in Madhya Pradesh, India
  Interventions: Behavioral: Smart phone based training
- In person training (Experimental): In person training for Headmasters to implement the Tobacco Free Teachers-Tobacco Free Society program in their schools in Madhya Pradesh, India
  Interventions: Behavioral: In person training

INTERVENTIONS:
Behavioral: Smart phone based training — The study team will acquaint headmasters with the Tobacco Free Teachers-Tobacco Free Society (TFT-TFS) program and the smartphone training app. Headmasters will receive six monthly trainings on smartphones, including brief videos followed by quizzes with feedback, discussion forums to promote peer learning, demonstration of techniques, and the ability to review the content as needed. Headmasters will implement TFT-TFS at monthly school meetings with teachers and parents. TFT-TFS consists of four program components: (1) six group discussions with teachers, (2) cessation support and referrals to government resources, (3) posting six thematic tobacco control posters in the school, and (4) implementing a school tobacco policy. These four components incorporate the program's six themes: Teachers as Role Models; Health Effects of Tobacco; Motivation to Quit Tobacco Use; Skills to Quit Tobacco and to Help Others Quit; Dealing with Withdrawal; and Maintenance and Celebration.
  Arms: Smart phone based training
Behavioral: In person training — Headmasters will receive three face-to-face trainings, each 60-75 minutes long and held at convenient locations. The study team will introduce headmasters to the TFT-TFS program and teach participants how to use paper-based materials. The trainings will encourage participants to discuss successes and come up with solutions to overcome challenges. Headmasters will implement TFT-TFS at monthly school meetings with teachers and parents. TFT-TFS consists of four program components: (1) 6 group discussions with teachers, (2) cessation support and referrals to government resources, (3) posting six thematic tobacco control posters in the school, and (4) implementing a school tobacco policy. These four components incorporate the program's six themes: Teachers as Role Models; Health Effects of Tobacco; Motivation to Quit Tobacco Use; Skills to Quit Tobacco and to Help Others Quit; Dealing with Withdrawal; and Maintenance and Celebration.
  Arms: In person training

SUMMARY:
This study aims to compare the implementation and effectiveness of the Tobacco-Free Teachers, Tobacco-Free Society (TFT-TFS) program when delivered through in-person training vs. a smartphone-based training model. Investigators will conduct a comparative effectiveness trial using a cluster-randomized design in which headmasters at schools in the Indian state of Madhya Pradesh (MP) will be trained in person or via a smartphone to deliver TFT-TFS in their schools. Schools will be randomly assigned to each training arm, and investigators will compare program effectiveness (tobacco use cessation), implementation outcomes, and program cost and reach.

DETAILED DESCRIPTION:
Tobacco-related deaths are rising rapidly in low and middle-income countries (LMICs). India's population is the second largest consumer of tobacco products in the world: 29% of the adult population uses smoked, smokeless, or both forms of tobacco, and around 1.2 million die each year from tobacco-related causes. Reducing tobacco-related deaths in LMICs will require large-scale implementation of evidence-based interventions (EBIs) that promote tobacco control. Currently, the implementation of tobacco control EBIs in LMICs relies on in-person training, which has inherent logistical challenges that limit the ability to scale up these programs. New training models are needed to ensure tobacco control EBIs can be implemented broadly, rapidly, and at low cost, especially in rural and under-resourced areas where tobacco use is prevalent.

The long-term goal is to identify effective, low-resource strategies to promote the broad-based implementation of tobacco control EBIs in LMICs. In India, school teachers are respected community leaders, role models, and an important channel for promoting tobacco control in schools and society. Investigators previously demonstrated the effectiveness of the Tobacco-Free Teachers, Tobacco-Free Society (TFT-TFS) program in a cluster-randomized study of schoolteachers in Bihar state, India. Tobacco use cessation rates were doubled among teachers in intervention schools compared to control schools, along with significant improvements in the adoption and implementation of tobacco control policies. As a critical next step in scaling up the TFT-TFS tobacco control EBI, investigators are focusing on expanding the training of those implementing the program in schools, i.e., school headmasters. The investigators will compare two models of TFT-TFS training of headmasters-in-person vs. smartphone-based-and the effect of each approach on TFT-TFS program implementation and effectiveness. India has the world's second-largest mobile phone user subscription base of 1.2 billion, with good penetration even in rural areas. The use of smartphones in educational settings is already pervasive in India, offering a readily available, low-cost strategy for expanding training of the TFT-TFS program. Training via smartphones can be delivered anytime and anywhere and allows flexibility and individualization of the learning experience through on-demand access to training content and virtual interactions among trainees. By delivering TFT-TFS training through smartphones, the program's potential reach can be multiplied over what can be achieved with in-person training.

Investigators will conduct a comparative effectiveness trial using a cluster-randomized design in which headmasters of schools in the Indian state of Madhya Pradesh (MP) will be randomly assigned to receive in-person training or training via smartphone for the TFT-TFS program. Once trained, headmasters in both groups will implement the TFT-TFS program within schools. Investigators will compare the training arms regarding program effectiveness (tobacco use cessation), implementation, cost, and reach.

ELIGIBILITY:
Inclusion Criteria:

All teachers and principals employed in schools in both study arms

Exclusion Criteria:

• None

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2040 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Tobacco use cessation among teachers | Baseline and Immediate post intervention
  Self-administered school personnel survey completed by teachers and principals. Based on the school personnel surveys, the investigators will assess self-report tobacco use at baseline and immediate post intervention and compare measures between the two arms to assess the effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Nagler, ScD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Healis Sekhsaria Institute for Public Health, Indore, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No